CLINICAL TRIAL: NCT05346068
Title: The Value of IVL Compared To OPN Non-Compliant Balloons for Treatment of RefractorY Coronary Lesions (VICTORY) Trial - A Randomized, Multicenter, Non-inferiority Comparison of Shockwave Intravascular Lithotripsy (IVL) and the OPN Non-compliant Balloon for Treatment of Calcified and Refractory Coronary Lesions
Brief Title: The Value of IVL Compared To OPN Non-Compliant Balloons for Treatment of RefractorY Coronary Lesions (VICTORY) Trial
Acronym: VICTORY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: Hôpital Fribourgeois (Other); Hamilton General Hospital (Unknown)
Responsible Party: Principal Investigator, Matthias Bossard, Co-Principal Investigator, Luzerner Kantonsspital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VICTORY Trial
Record Dates: First submitted 2022-03-31; First posted 2022-04-26 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Coronary Disease; Coronary Artery Disease; Calcific Coronary Arteriosclerosis; Stent Restenosis; Coronary Artery Calcification
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Prospective, randomized, multicenter, non-inferiority trial with blinded assessment of outcomes (PROBE design)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Device (Experimental)
  Interventions: Device: OPN™ NCB Super High Pressure PCI Balloon
- Control Device (Active Comparator)
  Interventions: Device: Shockwave™ C2 IVL Catheter

INTERVENTIONS:
Device: OPN™ NCB Super High Pressure PCI Balloon — In order to permit advancement of the studied medical devices - OPN™ NCB or Shockwave™ IVL balloon catheter - initial lesion preparation using small SCBs or NCBs (≤2mm) or rotablation (Boston Scientific, Marlborough, MA, United States) is allowed, but will be documented. This may be required in selected cases with very calcified and tight lesions.
  As per protocol, lesion preparation will be performed using either the super-high pressure PCI balloon OPN™ NCB or the Shockwave™ IVL balloon catheter according to random treatment assignment after matching the angiographic and/or OCT inclusion criteria.
  Following successful lesion preparation all patients will be treated with a latest generation durable polymer everolimus-eluting stent (Xience™ Sierra or Skypoint, Abbott Vascular Inc., Santa Clara, CA, United States) to allow comparison of stent expansion.
  Arms: Study Device
Device: Shockwave™ C2 IVL Catheter — In order to permit advancement of the studied medical devices - OPN™ NCB or Shockwave™ IVL balloon catheter - initial lesion preparation using small SCBs or NCBs (≤2mm) or rotablation (Boston Scientific, Marlborough, MA, United States) is allowed, but will be documented. This may be required in selected cases with very calcified and tight lesions.
  As per protocol, lesion preparation will be performed using either the super-high pressure PCI balloon OPN™ NCB or the Shockwave™ IVL balloon catheter according to random treatment assignment after matching the angiographic and/or OCT inclusion criteria.
  Following successful lesion preparation all patients will be treated with a latest generation durable polymer everolimus-eluting stent (Xience™ Sierra or Skypoint, Abbott Vascular Inc., Santa Clara, CA, United States) to allow comparison of stent expansion.
  Arms: Control Device

SUMMARY:
Percutaneous coronary intervention (PCI) with drug-eluting stent (DES) implantation has become the dominant treatment strategy for patients with acute and chronic coronary artery disease (CAD) requiring revascularization. Nonetheless, PCI with stent implantation has some limitations and especially patients with severely calcified coronary lesions (approximately 10-20% of all patients with CAD) have an elevated risk for adverse outcomes, including target lesion failure (TLF) and stent thrombosis (ST).

Several dedicated PCI devices have been developed for treatment of severely calcified lesions. Whereas especially two of them have shown promising results in smaller, prospective studies. First, the super high-pressure NC PCI balloon (OPN™ NC, SIS Medical AG, Frauenfeld, Switzerland) has been shown to represent an effective and safe device for lesion preparation. Second, the lately introduced Shockwave intravascular lithotripsy (IVL)™ balloon catheter (Shockwave Medical, Santa Clara, CA, USA) appears to be a safe and efficient alternative device for treatment of calcified coronary lesions. However, it remains unknown, if the OPN™ NC balloon is non-inferior to to IVL regarding lesion preparation and completeness of stent expansion in severely calcified lesions.

DETAILED DESCRIPTION:
To evaluate final stent expansion following a strategy of lesion preparation with either the Shockwave C2 IVL™ Catheter (Shockwave Medical Inc. Santa Clara, CA, United States) or a super high-Pressure NC PTCA Balloon (OPN™ NC; SIS Medical Distribution AG, Frauenfeld, Switzerland) in patients with heavily calcified coronary lesions undergoing coronary stent implantation.

To assess the safety of a strategy of using super high-pressure NC balloons compared to shockwave IVL™ for treatment of heavily calcified lesions, which are treated with a contemporary drug eluting stent.

Patients presenting with chronic or acute coronary artery disease and requiring PCI to a very calcified coronary artery lesion will either be randomized to preparation of that corresponding lesion using the control device (Shockwave™ IVL balloon catheter) or the study device (the super high-pressure NC PCI Balloon (OPN™ NC)).

The treatment of the calcified coronary lesion will be guided by use of intravascular imaging (optical coherence tomography, OCT).

Enrolled patients will undergo follow-up at 30 days, 1 year and 2 years

ELIGIBILITY:
Clinical inclusion criteria:

* Age ≥18 years and consentable;
* Acute or chronic coronary artery disease with ischemia related symptoms (e.g. angina) and/or evidence of myocardial ischemia (e.g. FFR/ iFR, CMR, SPECT or PET-CT);
* Angiographically-proven coronary artery disease;
* Lesions in non-target vessels requiring PCI may be treated either

  * prior to the study procedure if the procedure was unsuccessful or complicated; or
  * in the same session if feasible and safe for the patient, otherwise a staged PCI procedure for non-target vessels may be considered;
* Informed Consent signed by the subject.

Angiographic inclusion criteria:

* Single de novo target lesion stenosis of protected LMCA, or LAD, RCA or LCX (or of their branches) with*:

  * Stenosis of ≥70%;
  * Stenosis ≥50% and <70% (visually assessed) with evidence of ischemia via positive stress test, or fractional flow reserve value ≤0.80, or iFR <0.90 or IVUS minimum lumen area ≤4.0 mm²;
* The target vessel reference diameter must be ≥2.5 mm & ≤4.5mm;
* AND AT LEAST ONE OF THE FOLLOWING CRITERIA:

  * Evidence of calcification at the lesion site by angiography (Grade 3), with fluoroscopic radio-opacities noted without cardiac motion prior to contrast injection involving both sides of the arterial wall in at least one location and total length of calcium of at least 15 mm and extending partially into the target lesion,
  * AND/ OR by OCT, with presence of ≥270° calcium;
  * AND/ OR Prior attempt at PCI with inability to expand a balloon in target lesion.

Annotation: Only one lesion and vessel per randomized patient may be treated according to protocol and considered for the purpose of this study. The lesion considered for the study should represent the most calcified one.

The presence of any one of the following exclusion criteria will lead to the exclusion of the subject:

Exclusion criteria:

* Patient experienced an acute STEMI or cardiogenic shock related to an acute MI within 2 days prior to index procedure;
* Any comorbidity or condition which may reduce compliance with this protocol, including follow-up calls/ visits (e.g. advanced dementia);
* Any medical, geographic, and/or social factor making study participation impractical or precluding required follow-up.
* Patient is pregnant or nursing (a negative pregnancy test is required for women of child-bearing potential within 7 days prior to enrollment);
* Unable to take a P2Y12 inhibitor (i.e. clopidogrel, prasugrel, or ticagrelor) for at least 6 months;
* Patient has an allergy to imaging contrast media which cannot be adequately pre-medicated;
* Renal failure with an eGFR <30ml/min1.73m2;
* History of a stroke or transient ischemic attack (TIA) within 7 days, or any prior intracranial hemorrhage;
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within 6 months;
* Untreated pre-procedural hemoglobin <10g/dL or intention to refuse blood transfusions if one should become necessary;
* Patient has an allergy or intolerance to cobalt-chromium and/ or everolimus.
* Life expectancy of less than 1 year.

Angiographic exclusion criteria:

* Anatomy where the device or OCT catheter are unlikely to be delivered due to tortuosity or other characteristics;
* Target lesion is in a coronary artery bypass graft;
* Target lesion is an in-stent restenosis (ISR);
* Flow limiting target vessel thrombus (evident on angiography or OCT);
* Definite or possible thrombus (by angiography or intravascular imaging) in the target vessel;
* Evidence of aneurysm in target vessel within 10 mm of the target lesion.

Of note, only qualified physicians who are investigators or a sub-investigators for the trial will assess each individual´s eligibility criteria and take the final decision to include the subject in the trial (ICH GCP 4.3.1). This decision will be documented prior to the subject receiving the first intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Final stent expansion (in percentage, %) assessed by OCT | At index Procedure

SECONDARY OUTCOMES:
Acceptable stent expansion (>80%) assessed by OCT | At index Procedure
Optimal stent expansion (>90%) assessed by OCT | At index Procedure
Procedural success | At index Procedure
  defined as the achievement of angiographic success (residual stenosis of <30%, no flow-limiting dissection and/or no no-reflow) without any major adverse cardiac events (MACE), which is defined as cardiac death, target vessel related myocardial infarction, TIA/ stroke and repeat revascularization (PCI or CABG) up to 30 days
Strategy success | At index Procedure
  defined as procedural success using the assigned study device and stent, without requirement for lesion preparation with further devices (i.e. cross-over to the non-assigned study devices or cutting/ scoring balloons).

OTHER OUTCOMES:
Coronary perforations (Ellis grade III and/or cavity spilling) | At index Procedure
Persistent periprocedural vessel occlusion/MI | At index Procedure
Periprocedural ventricular tachycardia/fibrillation (VT/ VF) | At index Procedure
Contrast-induced nephropathy (CIN) | At index Procedure
Major bleeding (BARC 3-5) | At index Procedure, 30 days, 1 Year and 2 Years
Number of complementary lesion preparations with further devices (i.e. cutting or scoring balloons) or cross-over to the non-assigned study devices. | At index Procedure
Acute lumen gain | At index Procedure
  defined as minimal lumen diameter (MLD) post balloon angioplasty minus baseline MLD (mm) assessed by OCT
Frequency of calcium fracture/s (CF) at the site of maximum calcium | At index Procedure
Procedure duration | At index Procedure
Procedure radiation exposure | At index Procedure
Procedure contrast volume | At index Procedure
Major Adverse Cardiac Events (MACE) | At 30 days, 1 Year and 2 Years
  defined as cardiac death, target vessel related myocardial infarction, TIA/ stroke and repeat revascularization (PCI or CABG)
Target vessel revascularization (TVR) | At 30 days, 1 Year and 2 Years
  TVR is defined as any revascularization within the entire major coronary vessels proximal or distal to a target lesion including upstream and downstream side branches and the target lesion itself.
Target lesion revascularization (TLR) | At 30 days, 1 Year and 2 Years
  TLR is defined as any repeat percutaneous or surgical intervention due to a stenosis or occlusion within the stent or within the 5mm border proximal or distal to the stent.
Rate of new acute myocardial infarction (MI) (either NSTEMI/STEMI) | At 30 days, 1 Year and 2 Years
  MI is defined according to the Fourth Universal Definition of Myocardial Infarction. Peri-procedural MI is defined according to the Society of Coronary Angiography Interventions (SCAI) and Fourth Universal Definition of Myocardial Infarction definitions. SCAI criteria define peri-procedural MI as creatin kinase myocardial band measured (CK-MB) within 48 hours of the procedure elevated ≥10 times above the upper limit of normal (ULN), or ≥5 times ULN with development of new pathologic Q waves in 2 contiguous electrocardiographic leads or new left bundle branch block. In the absence of CK-MB measurements, post-procedural MI is defined as a troponin value ≥70 times ULN, or ≥35 times ULN with new pathologic Q waves or new left bundle branch block. The SCAI criteria to define peri-procedural MI were also used for patients with elevated cardiac enzymes at baseline.
Rate of Stent thrombosis (ST) | At 30 days, 1 Year and 2 Years
  According to ARC definition):
  1. Event certainty:
     * Definite: Acute coronary syndrome with angiographic or autopsy confirmations of stent thrombosis
     * Probable:
       i. Unexplained death within 30 days of stent implantation without autopsy. ii. Acute myocardial infarction in the territory of target vessel where stent was implanted but without angiographic confirmation.
     * Possible: Unexplained death after 30 days of stent implantation without autopsy.
  2. Time frame:
     * Early:
       i. Acute - during the procedure of stent implantation (PCI) ii. Sub-acute - within 30 days after PCI
     * Late: 1-12 months after stent implantation (up to 1 year)
     * Very late: After one year of stent implantation.
Rate of TIA or stroke | At 30 days, 1 Year and 2 Years
  Stroke requires the presence of acute focal or global neurological dysfunction caused by brain or retinal vascular injury due to primary hemorrhage or infarction. Symptoms or signs must persist >24 hours or when acute stroke is present on brain imaging (i.e. if there is an acute/subacute stroke documented by CT or MRI or at autopsy, the duration of symptoms/signs may be less than 24 hours).
  Global symptoms/signs are restricted to subarachnoid hemorrhage. Subarachnoid hemorrhage does not require focal neurological deficits, and the diagnosis is based on the clinical syndrome plus imaging as described below.
Rate of Cardiovascular death | At 30 days, 1 Year and 2 Years
  Cardiac death will be defined in accordance with the Academic Research Consortium (ARC) as any death due to a proximate cardiac cause (e.g. myocardial infarction, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause. All procedure-related deaths, including those related to concomitant treatment, will be classified as cardiac death.
Rate of all-cause death | At 30 days, 1 Year and 2 Years
  Includes death from any cause. The cause of death will be adjudicated.

CONTACTS AND LOCATIONS:
Locations (1):
- Luzerner Heart Centre, Lucerne, Switzerland

REFERENCES:
- [Background] Seiler T, Attinger-Toller A, Cioffi GM, Madanchi M, Teufer M, Wolfrum M, Moccetti F, Toggweiler S, Kobza R, Bossard M, Cuculi F. Treatment of In-Stent Restenosis Using a Dedicated Super High-Pressure Balloon. Cardiovasc Revasc Med. 2023 Jan;46:29-35. doi: 10.1016/j.carrev.2022.08.018. Epub 2022 Aug 20. PMID 36085285
- [Background] Pinilla-Echeverri N, Bossard M, Hillani A, Chavarria JA, Cioffi GM, Dutra G, Guerrero F, Madanchi M, Attinger A, Kossmann E, Sibbald M, Cuculi F, Sheth T. Treatment of Calcified Lesions Using a Dedicated Super-High Pressure Balloon: Multicenter Optical Coherence Tomography Registry. Cardiovasc Revasc Med. 2023 Jul;52:49-58. doi: 10.1016/j.carrev.2023.02.020. Epub 2023 Mar 2. PMID 36907698
- [Background] Cuculi F, Bossard M, Zasada W, Moccetti F, Voskuil M, Wolfrum M, Malinowski KP, Toggweiler S, Kobza R. Performing percutaneous coronary interventions with predilatation using non-compliant balloons at high-pressure versus conventional semi-compliant balloons: insights from two randomised studies using optical coherence tomography. Open Heart. 2020 Jan 23;7(1):e001204. doi: 10.1136/openhrt-2019-001204. eCollection 2020. PMID 32076567